CLINICAL TRIAL: NCT01399333
Title: Comparison of Meal Replacements Versus Protein Supplements and Utilizing the PDCAAS Method in the Bariatric Patient
Brief Title: Comparison of Meal Replacements Versus Protein Supplements and Utilizing the Protein Digestibility Corrected Amino Acid Score (PDCAAS) Method
Acronym: PDCAAS
Status: Unknown | Phase: Phase 4 | Type: Interventional
Last Known Status: Recruiting
Sponsor: Southeast Bariatrics, PA (Other)
Collaborators: University of North Carolina, Charlotte (Other)
Responsible Party: David C. Voellinger, MD, Southeast Bariatrics, an affiliate of Novant Medical Group
Allocation: Randomized | Model: Parallel | Masking: Single | Purpose: Screening
Other Study IDs: 10003
Record Dates: First submitted 2011-07-19; First posted 2011-07-21 (Estimated); Last update posted 2011-07-26 (Estimated); Status verified 2011-07

CONDITIONS: Protein Deficiency
Keywords: PDCAAS; Bariatric patient
MeSH Terms: conditions — Protein Deficiency

STUDY DESIGN:
Who Masked: Participant
Oversight: Data Monitoring Committee: No

ARMS (3):
- Group 1 (Active Comparator): full liquid diet utilizing meal replacements with PDCAAS of 1.0
  Interventions: Dietary Supplement: Group 1 Meal Replacement
- Group 2 (Active Comparator): full liquid diet utilizing protein supplements with PDCAAS of 0.5-0.99
  Interventions: Dietary Supplement: Group 2 Protein Supplement
- Group 3 (Active Comparator): full liquid diet utilizing protein supplement with a PDCAAS less than 0.5
  Interventions: Dietary Supplement: Group 3

INTERVENTIONS:
Dietary Supplement: Group 1 Meal Replacement — 4 weeks of utilizing Group 1 Meal Replacement 3-4 times daily, supplementing this protein product at each meal. As standard of care for the bariatric patient, they are required to get in 60-80 gms of protein daily
  Arms: Group 1
Dietary Supplement: Group 2 Protein Supplement — 4 weeks of utilizing Group 2 protein supplement 3-4 times daily, replacing this protein product at each meal. As standard of care for the bariatric patient, they are required to get in 60-80 gms of protein daily
  Arms: Group 2
Dietary Supplement: Group 3 — 4 weeks of utilizing Group 3 protein supplement 3-4 times daily, replacing this protein product at each meal. As standard of care for the bariatric patient, they are required to get in 60-80 gms of protein daily
  Arms: Group 3

SUMMARY:
The purpose of this research study is to compare the varying qualities of protein supplements utilizing the Protein Digestibility Corrected Amino Acid Score (PDCAAS) method and evaluating the clinical outcome related to protein stores and absorption.

DETAILED DESCRIPTION:
The PDCAAS has been adopted by the Food and Agricultural Organization (FAO) of the World Health Organization (WHO) and is currently recognized as the standard method to evaluate protein quality. This study will also examine patient tolerability, satiety, and satisfaction while using meal replacements versus protein supplements. This research study looks to gain knowledge on the varying qualities of protein and find the most effective protein supplement and/or meal replacement that provides increased patient compliance and promotes a healthy recovery.

ELIGIBILITY:
Inclusion Criteria:

* Persons that are scheduled to undergo the adjustable gastric banding (AGB) surgery utilizing the AP Lap-Band System.
* Not having any medical confounding factors as described in exclusion criteria.
* Willing to comply with food and exercise logs and comply with the full-liquid diet, both pre-and-post-operatively.

Exclusion Criteria:

* Persons who are not undergoing AGB surgery or are unwilling to comply with study methods or are medically not eligible.
* Taking diuretics
* Have been diagnosed with unstable diabetes, unstable neurologic conditions, unstable cardiac conditions or gastro-intestinal disorders, renal dysfunction, wounds, and autoimmune disorders that may increase protein needs.
* Uncontrolled gastrointestinal disease, such as Crohn's disease, diverticulitis, Celiac disease, or ulcerative colitis.
* Active malignancy
* Patients will also be excluded if pre-operative vitamin deficiencies are not corrected by surgery.

Ages: 18 Years to 65 Years | Sex: All | Healthy Volunteers: Yes
Age Groups: Adult, Older Adult
Enrollment: 60 (Estimated)
Dates: Start 2010-01; Primary Completion 2011-08 (Estimated); Study Completion 2012-01 (Estimated)

PRIMARY OUTCOMES:
Protein Absorption | 4 weeks
  protein stores and protein absorption per lab results collected at required visits

SECONDARY OUTCOMES:
Patient Compliance with Protein Supplement | 4 weeks
  Evaluate patient compliance with protein supplements during the required 4 week liquid diet phase, which include 2 weeks prior to surgery and 2 weeks after surgery.
Patient tolerability and satisfaction of protein supplement | 4 weeks
  Evaluate the patient's tolerability of the protein supplement, specifically assessing GI symptoms and satiety, as well as evaluating patient perceptions of satisfaction of the product and satiety.

CONTACTS AND LOCATIONS:
Overall Officials: David C Voellinger, MD, Principal Investigator — Southeast Bariatrics
Locations (1):
- Southeast Bariatrics, Charlotte, North Carolina, United States